CLINICAL TRIAL: NCT06840327
Title: Impact of VARIation of OXYdo-reduction Potential in Cardiac Surgery on Post-operative Outcome
Acronym: VARIOXY
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0523; ID-RCB (Other: 2025-A00118-41)
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Surgery; Extracorporeal Circulation
Keywords: extracorporeal circulation; cardiac surgery; biological markers; Redox balance; post-operative outcome
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surgical residue from incision surgery planned for surgery without additional incision; catheter samples: peripheral venous blood, central venous blood, peripheral arterial blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Scheduled cardiac surgery patients: Scheduled cardiac surgery patients undergoing bypass surgery with saphenous vein harvesting.
  Interventions: Other: Blood and tissue samples; Other: walking test

INTERVENTIONS:
Other: Blood and tissue samples — Blood samples will be taken from catheters placed for the purpose of surgery (arterial and venous catheters), or during routine venipunctures. (D-1 pre-op). Tissue samples will be taken from surgical waste generated by the surgery. They will therefore not require any additional incisions or surgical procedures.
Other: walking test — The study includes a walking test between D5 and D7.

SUMMARY:
Observational, prospective, monocentric study conducted in the cardiac surgery department about biological markers to predict the short-term outcome of heart surgery patients.

DETAILED DESCRIPTION:
At present, there are no biological markers to predict the short-term outcome of heart surgery patients. Redox balance, determined by the interaction between oxidants and reducers in tissues, is an essential parameter in the regulation of cellular functions. Cardiac surgery with extracorporeal circulation (CEC) induces major disturbances in this balance. In preliminary work, it was observed that the redox potential (Eg) varied with the introduction of CEC, and a persistent imbalance appeared to correlate with post-operative complications. It is believed that Eg potential could be a new biomarker of the post-operative outcome of major surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients over 18 years of age Scheduled cardiac surgery patients undergoing bypass surgery with saphenous vein harvesting.

Patients able to understand the protocol; Patients able to express non-opposition to participating in the study Patients affiliated to a social security system or equivalent.

Exclusion Criteria:

Emergency surgery patients. Pregnant or breast-feeding women. Patients deprived of their freedom or under legal protective measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing scheduled cardiac surgery under CEC for coronary bypass surgery with saphenous vein harvesting at Toulouse University Hospital
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Simplified Gravity Index | Day 7
  severity score used in intensive care to assess the risk of in-hospital mortality. Score from 0 to 163 points (0 is the best possible state of health / 163 is the worst possible state of health )

IPD SHARING:
Plan to Share IPD: No